CLINICAL TRIAL: NCT04382157
Title: Magnesium Replacement and Hyperglycemia After Kidney Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Trond Jenssen, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/842
Record Dates: First submitted 2020-05-03; First posted 2020-05-11 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Hypomagnesemia; Kidney Transplantation
Keywords: Oral glucose tolerance test; Magnesium hydroxide; hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mablet (Experimental): Mablet 360 mg. Twice daily for 4 weeks. If tolerated trice daily for following 20 weeks. Treatment for 24 weeks in total.
  Interventions: Drug: Mablet 360 mg
- Placebo (Placebo Comparator): Placebo. Twice daily for 4 weeks. If tolerated trice daily for following 20 weeks. Treatment for 24 weeks in total.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mablet 360 mg — Slow-released magnesium hydroxide
  Arms: Mablet
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The insulin receptor is dependent on magnesium and hypomagnesemia is associated with increased insulin resistance and decreased insulin secretion and action. Recent data suggest that hypomagnesemia may play a role in development of type 2 diabetes. Kidney transplantation patients have low plasma magnesium levels, partly due to treatment with calcineurin inhibitors. However, the role of magnesium in the development of post-transplant diabetes mellitus (PTDM) is unclear.

The present study addresses, whether hypomagnesemia is feasible to reverse by oral administration of magnesium.

The investigators wish to investigate whether oral magnesium supplementation is sufficient to increase magnesium levels in kidney transplant recipients, and if supplementation improves glycemic parameters as measured by an oral glucose tolerance test (OGTT).

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients more than one year after transplantation
* Hypomagnesemia (< 0.7 mmol/L)
* Age ≥ 18 years and able to give written informed consent

Exclusion Criteria:

* Current treatment with magnesium containing medication or supplements
* Current medical treatment for diabetes
* Conditions impairing magnesium absorption from the gastrointestinal tract (e.g. short bowel syndrome, chronic pancreatitis)
* Subjects with primary non-graft function and subjects with need of dialysis therapy >2 months or graftectomy at any time point after transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Magnesium retension at loading test | 24 weeks
  Difference in magnesium retension at magnesium loading test between before and after oral treatment. Retension defined as percentage of magnesium retained from intravenous magnesium sulphate.

SECONDARY OUTCOMES:
Plasma glucose (mmol/L) | Baseline (Before magnesium loading tests)
  Change of fasting plasma glucose (mmol/L) between start and the end of supplementation.
Insulin (mg/kg/min) | 2 hours oral glucose tolerance test
  Change of insulin (mg/kg/min) in OGTT (after 2 hours) between start and the end of supplementation.
C-peptide (nmol/L) | 2 hours oral glucose tolerance test
  Change of C-peptide (nmol/L) in OGTT (after 2 hours) between start and the end of supplementation.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No